CLINICAL TRIAL: NCT05752383
Title: The Clinical and Hemodynamic Course of Cardiogenic Shocks Hospitalized in Critical Care
Acronym: HEMOCARD
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2022_843_0132
Record Dates: First submitted 2023-01-24; First posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic Shock; vaso-inotropic score
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiogenic shock is a frequent reason for hospitalization in critical care units, with high mortality (50%). Several French registries have been created to improve knowledge of the prognostic factors of cardiogenic shock. In recent years, temporary mechanical circulatory support has become more important in cardiogenic shock. The monitoring of catecholamines is also performed with a global score: the vaso-inotropic score. The purpose of our study is to consider using these new data and techniques to create a cohort of cardiogenic shock within our critical care unit.

This observational study is based on clinical, biological, and hemodynamic data recorded during the ICU stay of patients for cardiogenic shock.

The primary endpoint is the relationship between the hemodynamic evolution of cardiogenic shock and in-hospital mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in ICU for cardiogenic shock
* Patient with cardiogenic shock as defined by the FRENSCHOCK2 study criteria

Exclusion Criteria:

* Patient with cardiogenic shock in the context of septic shock and hemorrhagic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients hospitalized in ICU for cardiogenic shock
  * Patient with cardiogenic shock as defined by the FRENSCHOCK2 study criteria
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-24 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of in-hospital mortality after cardiogenic shock | 5 years
Vaso-inotropic score after cardiogenic shock | 5 years
  vasoactive-inotropic score (VIS) Maximal VIS (VISmax) is calculated using the highest doses of vasoactive and inotropic medications administered.
  VISmax categories: 0-5, >5-15, >15-30, >30-45, and >45 points.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, France